CLINICAL TRIAL: NCT00312403
Title: Polymorphisms in the Human Matrix Metalloproteinase Genes MMP1, MMP3, and MMP9: Genetic Risk Factors of Primary Open Angle Glaucoma?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gabriele Fuchsjaeger-Mayrl, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OPHT-300505
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Glaucoma
Keywords: Glaucoma; Gene Polymorphism; Metalloproteinase
MeSH Terms: conditions — Glaucoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Patients with primary open angle glaucoma
  Interventions: Procedure: Blood Sample
- 2 (Other): Age- and sex-matched control subjects
  Interventions: Procedure: Blood Sample

INTERVENTIONS:
Procedure: Blood Sample — A single venous blood sample will be taken (10 ml).

SUMMARY:
Matrix metalloproteinases (MMPs) fulfill diverse important molecular functions and play pivotal roles in development, tissue morphogenesis, repair, aging, and inflammatory processes. MMPs are also important disease modulating factors, such as cancer, cardiovascular disease, rheumatoid arthritis or macular degeneration. Functional genetic variants have been described to fine-tune MMP activities at the gene transcriptional level and have been associated with increased genetic risk of e.g. arteriosclerosis or cancer. MMPs are also assumed to play a major role in the remodeling of the extracellular matrix (ECM) in the optic nerve head during glaucomatous optic neuropathy. MMP-1, MMP-3 and MMP-9 have been shown to be up-regulated in a variety of animal models of glaucoma. Here, we study three promoter SNPs within the genes encoding three members of the MMP family. By assessing the prevalence of genetic variants associated with either increased/decreased enzyme activity, we will (i) estimate their contribution to the genetic risk of developing primary open angle glaucoma (POAG) and (ii) investigate the potential role of MMPs in the functional pathology of POAG.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 39 years
* Primary open angle glaucoma as evidenced from characteristic visual field loss and optic disc cupping (POAG group)
* Healthy subjects matched by age, sex and ethnicity to the POAG patients group (control group)

Exclusion Criteria:

* Exfoliation glaucoma, pigmentary glaucoma
* History of acute angle closure

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2005-11; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Genotyping results and putatively associated odds with occurence of primary open angle glaucoma. | 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjaeger-Mayrl, M.D., Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria